CLINICAL TRIAL: NCT07206303
Title: The Effects of Bifidobacterium-based Probiotics in Reducing Blood Pressure in Middle-aged Chinese With Hypertension: a Single-term Feasibility Pilot Study
Brief Title: The Effects of Bifidobacterium-based Probiotics in Reducing Blood Pressure in Middle-aged Chinese With Hypertension
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Gary Kui Kai LAU, Clinical Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GL202401
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Hypertension
Keywords: hypertension; Bifidobacterium; probiotics
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 30 recruited participants receiving commercially available probiotics supplements (Experimental): 30 community-dwelling, middle-aged Hong Kong Chinese (15 men and 15 women) with hypertension according to ACC/AHA guidelines (SBP ≥130 mm Hg) who are not taking antihypertensive agents and are free of symptomatic cardiovascular or cerebrovascular diseases will be recruited in this study. Participants will be recruited via our outreach promotion program or social media and recruitment posters will be distributed physically or posted online.
  Interventions: Biological: Bifidobacterium probiotics supplementation

INTERVENTIONS:
Biological: Bifidobacterium probiotics supplementation — The 10-week research period consists of one prescreening and baseline visit (week -1) and two follow-up visits (week 5 (±7days) and week 10 (±7days)). The participants will be instructed to fast overnight before their visits in the mornings of week -1 and week 10.
  The measurements will include documentation of personal and demographic information; three consecutive clinic BP readings; 24-hour ambulatory BP monitoring; a 3-day diet diary to monitor consistency of dietary intake; collection of fecal samples and blood samples for analysis of GM composition and biomarkers, respectively at baseline, and week 5 and 10.
  Only participants who are able to provide all the required data and samples within 7 days after the prescreening and baseline visit (week -1) will be eligible to receive the Bifidobacterium supplementation with 20 billion cfu once a day for 10 weeks. They will be instructed to mix the probiotics with water and consume with their dinner.

SUMMARY:
The primary objective of this study is to investigate if a Bifidobacterium-based probiotic intervention would reduce clinic systolic BP in untreated middle-aged Chinese men and women with hypertension according to ACC/AHA guidelines (SBP ≥130 mm Hg) after 10 weeks of treatment. The investigators anticipate that this feasibility study will provide rationale to conduct a larger randomized clinical trial and preliminary data to estimate the power/ sample size of a larger RCT.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate if a Bifidobacterium-based probiotic intervention would reduce clinic systolic BP in untreated middle-aged Chinese men and women with hypertension according to ACC/AHA guidelines (SBP ≥130 mm Hg) after 10 weeks of treatment. The investigators anticipate that this feasibility study will provide rationale to conduct a larger randomized clinical trial and preliminary data to estimate the power/ sample size of a larger RCT.

The four independent but interrelated objectives of this study include:

1. To investigate if oral administration of Bifidobacterium-based probiotic intervention will reduce clinic SBP and DBP from baseline to the end of treatment.
2. To observe changes in 24-hour mean, daytime and nighttime SBP and DBP assessed by 24-hour ambulatory BP monitoring from baseline to the end of treatment.
3. To evaluate the impact of probiotics intervention on gut microbiome (GM) composition and functions characterized by shotgun metagenomic sequencing of stool.
4. To explore potential underlying mechanisms of Bifidobacterium-based probiotics on lowering BP by assessing serum proinflammatory and oxidative stress markers and circulating GM-derived metabolites, including SCFAs and GABA.

Additionally, the investigators will conduct sex-stratified analysis to explore potential sex differences in BP lowering response to the intervention since sex-linked differences in the initiation and progression of hypertension pathology are well-established, and the investigators recently reported that association between GM and hypertension is also sex-linked.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, aged 40-65 years old.
* Chinese residing in Hong Kong.
* Clinic SBP ≥130mmHg according to screening measurement at baseline.
* Untreated or not on antihypertensive medications within 4 weeks.
* Able to provide informed consent.

Exclusion Criteria:

* Clinic SBP >165mmHg according to screening measurement at baseline
* Known history of diabetes, coronary artery disease, stroke, peripheral artery disease, malignancy or chronic kidney disease
* Known history of gastrointestinal disorders including inflammatory bowel disease, irritable bowel syndrome, Helicobacter pylori infection, liver cirrhosis or long-term use of proton pump inhibitors.
* Known increased risk of infection due to endovascular or rheumatic heart disease, endovascular grafts, congenital heart defects, endocarditis, mechanical heart valves, and permanent endovascular devices including permanent (not temporary) hemodialysis catheters, pacemakers, or defibrillators.
* Known secondary causes of hypertension.
* Currently taking omega-3 fatty acid supplements, probiotics, antibiotics, rifaximin, steroids, and antihypertensive agents within 4 weeks.
* Currently taking anti-oxidant vitamins within 6 months.
* Recent travel to tropical areas within 6 months.
* Recent bariatric surgery, hepatic resection, intestinal resection/colectomy, or any surgery within 3 months before the study.
* Identified higher susceptibility to infections caused by immunosuppression, such as a history of organ or hematopoietic stem cell (HSCs) transplant, neutropenia (ANC <500 cells/µl), HIV, and CD4 <200 cells/µl.
* Known allergies to any components of commercially-available probiotic supplements.
* Women who are pregnant, or intending to become pregnant, or lactation.
* Intending to participate or have participated in a clinical or nutritional intervention study in the last 30 days before study enrolment.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mean seated clinic systolic blood pressure (SBP) | During clinical visits at: - Baseline (a week prior to treatment), - Week 5 of treatment - Week 10 of treatment (end of treatment)
  Three consecutive BP measurements will be assessed using an automatic BP monitor, Microlife BP A200 AFIB (Microlife, Taiwan). Prior to taking BP measurements, participants will be instructed to sit and rest for at least five minutes. Participants will be advised to maintain an upright posture, with their arms positioned at heart level and palms facing upwards. Additionally, they will be advised to refrain from speaking during process. The average of three BP measurements will be taken to minimize random error.

SECONDARY OUTCOMES:
Mean seated clinic diastolic blood pressure (DBP) | During clinical visits at: - Baseline (a week prior to treatment), - Week 5 of treatment - Week 10 of treatment (end of treatment)
  Three consecutive BP measurements will be assessed using an automatic BP monitor, Microlife BP A200 AFIB (Microlife, Taiwan). Prior to taking BP measurements, participants will be instructed to sit and rest for at least five minutes. Participants will be advised to maintain an upright posture, with their arms positioned at heart level and palms facing upwards. Additionally, they will be advised to refrain from speaking during process. The average of three BP measurements will be taken to minimize random error.
Mean 24-hour ambulatory SBP | During clinical visits at: - Baseline (a week prior to treatment), - Week 10 of treatment (end of treatment)
  A calibrated ambulatory BP monitoring device, TM-2441 (A&D Medical, Japan) will be fitted onto the participants, with the BP cuff placed on their non-dominant arm to record the 24-hour ambulatory BP. The BP will be measured every 30 minutes from 6 am to 10 pm and then every 60 minutes from 10 pm to 6 am.
Gut microbiome composition and functions | During clinical visits at: - Baseline (a week prior to treatment), - Week 10 of treatment (end of treatment)
  Stool GM sequencing will be performed to compare GM abundance before and after probiotics intervention. This will enable metagenomic assembly community profiling and functional profiling, while facilitating the identification of presented taxa, their abundance, biochemical potential, and other relevant information. Other GM species that may be associated with hypertension could also be identified and provide valuable insights for the development of future GM-based intervention strategies. A set of OMNIgene-OMR205 kits (DNA Genotek, Canada) will be utilized for the collection and stabilization of gut microbial DNA and RNA, facilitating the profiling of gut microbiomes. We will also inquire about the participants' bowel habit concurrently, utilizing the Bristol Stool Chart as reference.
Plasma levels of gut microbiome-derived metabolites, short-chain fatty acids (SCFA) and gamma amino butyric acids (GABA) | During clinical visits at: - Baseline (a week prior to treatment), - Week 10 of treatment (end of treatment)
  The level of SCFAs in blood sample will be detected by a two-steps analysis: the blood sample will be first derivatized by 1-propanol/pyridine (3:2, v: v) and propyl chloroformate followed by the quantification using 7890B gas chromatography-mass spectrometry after centrifugation of blood.
Serum levels of proinflammatory and oxidative stress markers | During clinical visits at: - Baseline (a week prior to treatment), - Week 10 of treatment (end of treatment)
  Various inflammatory markers, including IL-1, IL-6, IL-8, TNF-α, IL-10 will be assessed using LEGENDplex™ 13-plex pro-inflammatory cytokine panel (BioLegend Inc., USA). Damages caused by radicals or excessive oxidants will be measured in the blood. DNA/RNA damage will be assessed by 8-Hydroxygaunaosine (8-OHG) or detecting the general DNA damage via comet assay. Lipid damage will be assessed by measuring malondialdehyde (MDA) levels and protein modification will be assessed by measuring the levels of advanced glycation end products (AGE).
  A portion of every blood sample will also be collected and preserved in a PAXgene Blood RNA tube manufactured by QIAGEN in Germany. This tube enables the extraction and purification of intracellular RNA for subsequent molecular diagnostic testing.
Sex differences in BP reduction after the intervention | Demographics to be collected during baseline visit.

CONTACTS AND LOCATIONS:
Overall Officials: Gary KK Lau, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chumpitazi BP, Self MM, Czyzewski DI, Cejka S, Swank PR, Shulman RJ. Bristol Stool Form Scale reliability and agreement decreases when determining Rome III stool form designations. Neurogastroenterol Motil. 2016 Mar;28(3):443-8. doi: 10.1111/nmo.12738. Epub 2015 Dec 21. PMID 26690980
- [Background] Kolodziejczyk AA, Zheng D, Elinav E. Diet-microbiota interactions and personalized nutrition. Nat Rev Microbiol. 2019 Dec;17(12):742-753. doi: 10.1038/s41579-019-0256-8. Epub 2019 Sep 20. PMID 31541197
- [Background] Azzi A. Oxidative Stress: What Is It? Can It Be Measured? Where Is It Located? Can It Be Good or Bad? Can It Be Prevented? Can It Be Cured? Antioxidants (Basel). 2022 Jul 23;11(8):1431. doi: 10.3390/antiox11081431. PMID 35892633
- [Background] Okita Y, Nakamura H, Kouda K, Takahashi I, Takaoka T, Kimura M, Sugiura T. Effects of vegetable containing gamma-aminobutyric acid on the cardiac autonomic nervous system in healthy young people. J Physiol Anthropol. 2009;28(3):101-7. doi: 10.2114/jpa2.28.101. PMID 19483370
- [Background] Hayakawa K, Kimura M, Kamata K. Mechanism underlying gamma-aminobutyric acid-induced antihypertensive effect in spontaneously hypertensive rats. Eur J Pharmacol. 2002 Mar 1;438(1-2):107-13. doi: 10.1016/s0014-2999(02)01294-3. PMID 11906718
- [Background] Verhaar BJH, Prodan A, Nieuwdorp M, Muller M. Gut Microbiota in Hypertension and Atherosclerosis: A Review. Nutrients. 2020 Sep 29;12(10):2982. doi: 10.3390/nu12102982. PMID 33003455
- [Background] Zheng X, Qiu Y, Zhong W, Baxter S, Su M, Li Q, Xie G, Ore BM, Qiao S, Spencer MD, Zeisel SH, Zhou Z, Zhao A, Jia W. A targeted metabolomic protocol for short-chain fatty acids and branched-chain amino acids. Metabolomics. 2013 Aug 1;9(4):818-827. doi: 10.1007/s11306-013-0500-6. PMID 23997757
- [Background] Virwani PD, Qian G, Hsu MSS, Pijarnvanit TKKTS, Cheung CN, Chow YH, Tang LK, Tse YH, Xian JW, Lam SS, Lee CPI, Lo CCW, Liu RKC, Ho TL, Chow BY, Leung KS, Tsang HW, Lo EKK, Tung KTS, Chung SK, Yuen MF, Leung SY, Ip P, Hung IF, Louie JCY, El-Nezami H, Ho JWK, Lau KK. Sex Differences in Association Between Gut Microbiome and Essential Hypertension Based on Ambulatory Blood Pressure Monitoring. Hypertension. 2023 Jun;80(6):1331-1342. doi: 10.1161/HYPERTENSIONAHA.122.20752. Epub 2023 Apr 19. PMID 37073724
- [Background] Gerdts E, Sudano I, Brouwers S, Borghi C, Bruno RM, Ceconi C, Cornelissen V, Dievart F, Ferrini M, Kahan T, Lochen ML, Maas AHEM, Mahfoud F, Mihailidou AS, Moholdt T, Parati G, de Simone G. Sex differences in arterial hypertension. Eur Heart J. 2022 Dec 7;43(46):4777-4788. doi: 10.1093/eurheartj/ehac470. PMID 36136303
- [Background] Lau RI, Su Q, Lau ISF, Ching JYL, Wong MCS, Lau LHS, Tun HM, Mok CKP, Chau SWH, Tse YK, Cheung CP, Li MKT, Yeung GTY, Cheong PK, Chan FKL, Ng SC. A synbiotic preparation (SIM01) for post-acute COVID-19 syndrome in Hong Kong (RECOVERY): a randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2024 Mar;24(3):256-265. doi: 10.1016/S1473-3099(23)00685-0. Epub 2023 Dec 7. PMID 38071990
- [Background] Su Q, Liu Q, Zhang L, Xu Z, Liu C, Lu W, Ching JY, Li A, Mak JWY, Lui GCY, Ng SSS, Chow KM, Hui DS, Chan PK, Chan FKL, Ng SC. Antibiotics and probiotics impact gut antimicrobial resistance gene reservoir in COVID-19 patients. Gut Microbes. 2022 Jan-Dec;14(1):2128603. doi: 10.1080/19490976.2022.2128603. PMID 36201636
- [Background] Zhang L, Xu Z, Mak JWY, Chow KM, Lui G, Li TCM, Wong CK, Chan PKS, Ching JYL, Fujiwara Y, Chan FKL, Ng SC. Gut microbiota-derived synbiotic formula (SIM01) as a novel adjuvant therapy for COVID-19: An open-label pilot study. J Gastroenterol Hepatol. 2022 May;37(5):823-831. doi: 10.1111/jgh.15796. Epub 2022 Mar 2. PMID 35170078
- [Background] Chang BJ, Park SU, Jang YS, Ko SH, Joo NM, Kim SI, Kim CH, Chang DK. Effect of functional yogurt NY-YP901 in improving the trait of metabolic syndrome. Eur J Clin Nutr. 2011 Nov;65(11):1250-5. doi: 10.1038/ejcn.2011.115. Epub 2011 Jun 22. PMID 21697819
- [Background] Savard P, Lamarche B, Paradis ME, Thiboutot H, Laurin E, Roy D. Impact of Bifidobacterium animalis subsp. lactis BB-12 and, Lactobacillus acidophilus LA-5-containing yoghurt, on fecal bacterial counts of healthy adults. Int J Food Microbiol. 2011 Sep 1;149(1):50-7. doi: 10.1016/j.ijfoodmicro.2010.12.026. Epub 2011 Jan 15. PMID 21296446
- [Background] Agerholm-Larsen L, Raben A, Haulrik N, Hansen AS, Manders M, Astrup A. Effect of 8 week intake of probiotic milk products on risk factors for cardiovascular diseases. Eur J Clin Nutr. 2000 Apr;54(4):288-97. doi: 10.1038/sj.ejcn.1600937. PMID 10745279
- [Background] Usinger L, Ibsen H, Linneberg A, Azizi M, Flambard B, Jensen LT. Human in vivo study of the renin-angiotensin-aldosterone system and the sympathetic activity after 8 weeks daily intake of fermented milk. Clin Physiol Funct Imaging. 2010 Mar;30(2):162-8. doi: 10.1111/j.1475-097X.2009.00921.x. Epub 2010 Jan 26. PMID 20113315
- [Background] van der Zander K, Jakel M, Bianco V, Koning MM. Fermented lactotripeptides-containing milk lowers daytime blood pressure in high normal-to-mild hypertensive subjects. J Hum Hypertens. 2008 Nov;22(11):804-6. doi: 10.1038/jhh.2008.59. Epub 2008 Jun 5. PMID 18528405
- [Background] Sano J, Ohki K, Higuchi T, Aihara K, Mizuno S, Kajimoto O, Nakagawa S, Kajimoto Y, Nakamura Y. Effect of casein hydrolysate, prepared with protease derived from Aspergillus oryzae, on subjects with high-normal blood pressure or mild hypertension. J Med Food. 2005 Winter;8(4):423-30. doi: 10.1089/jmf.2005.8.423. PMID 16379551
- [Background] Jauhiainen T, Vapaatalo H, Poussa T, Kyronpalo S, Rasmussen M, Korpela R. Lactobacillus helveticus fermented milk lowers blood pressure in hypertensive subjects in 24-h ambulatory blood pressure measurement. Am J Hypertens. 2005 Dec;18(12 Pt 1):1600-5. doi: 10.1016/j.amjhyper.2005.06.006. PMID 16364832
- [Background] Aihara K, Kajimoto O, Hirata H, Takahashi R, Nakamura Y. Effect of powdered fermented milk with Lactobacillus helveticus on subjects with high-normal blood pressure or mild hypertension. J Am Coll Nutr. 2005 Aug;24(4):257-65. doi: 10.1080/07315724.2005.10719473. PMID 16093403
- [Background] Mizuno S, Matsuura K, Gotou T, Nishimura S, Kajimoto O, Yabune M, Kajimoto Y, Yamamoto N. Antihypertensive effect of casein hydrolysate in a placebo-controlled study in subjects with high-normal blood pressure and mild hypertension. Br J Nutr. 2005 Jul;94(1):84-91. doi: 10.1079/bjn20051422. PMID 16115337
- [Background] Hata Y, Yamamoto M, Ohni M, Nakajima K, Nakamura Y, Takano T. A placebo-controlled study of the effect of sour milk on blood pressure in hypertensive subjects. Am J Clin Nutr. 1996 Nov;64(5):767-71. doi: 10.1093/ajcn/64.5.767. PMID 8901799
- [Background] Tuomilehto J, Lindstrom J, Hyyrynen J, Korpela R, Karhunen ML, Mikkola L, Jauhiainen T, Seppo L, Nissinen A. Effect of ingesting sour milk fermented using Lactobacillus helveticus bacteria producing tripeptides on blood pressure in subjects with mild hypertension. J Hum Hypertens. 2004 Nov;18(11):795-802. doi: 10.1038/sj.jhh.1001745. PMID 15175633
- [Background] Inoue K, Shirai T, Ochiai H, Kasao M, Hayakawa K, Kimura M, Sansawa H. Blood-pressure-lowering effect of a novel fermented milk containing gamma-aminobutyric acid (GABA) in mild hypertensives. Eur J Clin Nutr. 2003 Mar;57(3):490-5. doi: 10.1038/sj.ejcn.1601555. PMID 12627188
- [Background] Wong MCS, Zhang L, Ching JYL, Mak JWY, Huang J, Wang S, Mok CKP, Wong A, Chiu OL, Fung YT, Cheong PK, Tun HM, Ng SC, Chan FKL. Effects of Gut Microbiome Modulation on Reducing Adverse Health Outcomes among Elderly and Diabetes Patients during the COVID-19 Pandemic: A Randomised, Double-Blind, Placebo-Controlled Trial (IMPACT Study). Nutrients. 2023 Apr 20;15(8):1982. doi: 10.3390/nu15081982. PMID 37111201
- [Background] Shimada M, Hasegawa T, Nishimura C, Kan H, Kanno T, Nakamura T, Matsubayashi T. Anti-hypertensive effect of gamma-aminobutyric acid (GABA)-rich Chlorella on high-normal blood pressure and borderline hypertension in placebo-controlled double blind study. Clin Exp Hypertens. 2009 Jun;31(4):342-54. doi: 10.1080/10641960902977908. PMID 19811362
- [Background] Ma P, Li T, Ji F, Wang H, Pang J. Effect of GABA on blood pressure and blood dynamics of anesthetic rats. Int J Clin Exp Med. 2015 Aug 15;8(8):14296-302. eCollection 2015. PMID 26550413
- [Background] Duranti S, Ruiz L, Lugli GA, Tames H, Milani C, Mancabelli L, Mancino W, Longhi G, Carnevali L, Sgoifo A, Margolles A, Ventura M, Ruas-Madiedo P, Turroni F. Bifidobacterium adolescentis as a key member of the human gut microbiota in the production of GABA. Sci Rep. 2020 Aug 24;10(1):14112. doi: 10.1038/s41598-020-70986-z. PMID 32839473
- [Background] Li Y, He L, Zhao Q, Bo T. Microbial and metabolic profiles of bronchopulmonary dysplasia and therapeutic effects of potential probiotics Limosilactobacillus reuteri and Bifidobacterium bifidum. J Appl Microbiol. 2022 Aug;133(2):908-921. doi: 10.1111/jam.15602. Epub 2022 May 16. PMID 35488863
- [Background] Lu W, Wang Y, Fang Z, Wang H, Zhu J, Zhai Q, Zhao J, Zhang H, Chen W. Bifidobacterium longum CCFM752 prevented hypertension and aortic lesion, improved antioxidative ability, and regulated the gut microbiome in spontaneously hypertensive rats. Food Funct. 2022 Jun 6;13(11):6373-6386. doi: 10.1039/d1fo04446j. PMID 35615892
- [Background] Averina OV, Kovtun AS, Mavletova DA, Ziganshin RH, Danilenko VN, Mihaylova D, Blazheva D, Slavchev A, Brazkova M, Ibrahim SA, Krastanov A. Oxidative Stress Response of Probiotic Strain Bifidobacterium longum subsp. longum GT15. Foods. 2023 Sep 7;12(18):3356. doi: 10.3390/foods12183356. PMID 37761064
- [Background] Fan L, Qi Y, Qu S, Chen X, Li A, Hendi M, Xu C, Wang L, Hou T, Si J, Chen S. B. adolescentis ameliorates chronic colitis by regulating Treg/Th2 response and gut microbiota remodeling. Gut Microbes. 2021 Jan-Dec;13(1):1-17. doi: 10.1080/19490976.2020.1826746. PMID 33557671
- [Background] Chen S, Chen L, Qi Y, Xu J, Ge Q, Fan Y, Chen D, Zhang Y, Wang L, Hou T, Yang X, Xi Y, Si J, Kang L, Wang L. Bifidobacterium adolescentis regulates catalase activity and host metabolism and improves healthspan and lifespan in multiple species. Nat Aging. 2021 Nov;1(11):991-1001. doi: 10.1038/s43587-021-00129-0. Epub 2021 Nov 16. PMID 37118342
- [Background] Bai B, Yang Y, Wang Q, Li M, Tian C, Liu Y, Aung LHH, Li PF, Yu T, Chu XM. NLRP3 inflammasome in endothelial dysfunction. Cell Death Dis. 2020 Sep 18;11(9):776. doi: 10.1038/s41419-020-02985-x. PMID 32948742
- [Background] Sun HJ, Ren XS, Xiong XQ, Chen YZ, Zhao MX, Wang JJ, Zhou YB, Han Y, Chen Q, Li YH, Kang YM, Zhu GQ. NLRP3 inflammasome activation contributes to VSMC phenotypic transformation and proliferation in hypertension. Cell Death Dis. 2017 Oct 5;8(10):e3074. doi: 10.1038/cddis.2017.470. PMID 28981106
- [Background] Rodrigo R, Gonzalez J, Paoletto F. The role of oxidative stress in the pathophysiology of hypertension. Hypertens Res. 2011 Apr;34(4):431-40. doi: 10.1038/hr.2010.264. Epub 2011 Jan 13. PMID 21228777
- [Background] Montezano AC, Touyz RM. Oxidative stress, Noxs, and hypertension: experimental evidence and clinical controversies. Ann Med. 2012 Jun;44 Suppl 1:S2-16. doi: 10.3109/07853890.2011.653393. PMID 22713144
- [Background] Zhang Z, Zhao L, Zhou X, Meng X, Zhou X. Role of inflammation, immunity, and oxidative stress in hypertension: New insights and potential therapeutic targets. Front Immunol. 2023 Jan 10;13:1098725. doi: 10.3389/fimmu.2022.1098725. eCollection 2022. PMID 36703963
- [Background] Joseph TA, Pe'er I. An Introduction to Whole-Metagenome Shotgun Sequencing Studies. Methods Mol Biol. 2021;2243:107-122. doi: 10.1007/978-1-0716-1103-6_6. PMID 33606255
- [Background] Zhao TX, Zhang L, Zhou N, Sun DS, Xie JH, Xu SK. Long-term use of probiotics for the management of office and ambulatory blood pressure: A systematic review and meta-analysis of randomized, controlled trials. Food Sci Nutr. 2022 Sep 20;11(1):101-113. doi: 10.1002/fsn3.3069. eCollection 2023 Jan. PMID 36655084
- [Background] Khalesi S, Sun J, Buys N, Jayasinghe R. Effect of probiotics on blood pressure: a systematic review and meta-analysis of randomized, controlled trials. Hypertension. 2014 Oct;64(4):897-903. doi: 10.1161/HYPERTENSIONAHA.114.03469. Epub 2014 Jul 21. PMID 25047574
- [Background] Dong JY, Szeto IM, Makinen K, Gao Q, Wang J, Qin LQ, Zhao Y. Effect of probiotic fermented milk on blood pressure: a meta-analysis of randomised controlled trials. Br J Nutr. 2013 Oct;110(7):1188-94. doi: 10.1017/S0007114513001712. Epub 2013 Jul 3. PMID 23823502
- [Background] Li J, Zhao F, Wang Y, Chen J, Tao J, Tian G, Wu S, Liu W, Cui Q, Geng B, Zhang W, Weldon R, Auguste K, Yang L, Liu X, Chen L, Yang X, Zhu B, Cai J. Gut microbiota dysbiosis contributes to the development of hypertension. Microbiome. 2017 Feb 1;5(1):14. doi: 10.1186/s40168-016-0222-x. PMID 28143587
- [Background] Muralitharan RR, Jama HA, Xie L, Peh A, Snelson M, Marques FZ. Microbial Peer Pressure: The Role of the Gut Microbiota in Hypertension and Its Complications. Hypertension. 2020 Dec;76(6):1674-1687. doi: 10.1161/HYPERTENSIONAHA.120.14473. Epub 2020 Oct 5. PMID 33012206
- [Background] Hamrahian SM, Maarouf OH, Fulop T. A Critical Review of Medication Adherence in Hypertension: Barriers and Facilitators Clinicians Should Consider. Patient Prefer Adherence. 2022 Oct 7;16:2749-2757. doi: 10.2147/PPA.S368784. eCollection 2022. PMID 36237983